CLINICAL TRIAL: NCT04709497
Title: Surgery for Primary Congenital Glaucoma in Neonates:Randomized Controlled Study.
Brief Title: Surgery for Primary Congenital Glaucoma in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Lecturer of ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Viscotrabeculotomy VI
Record Dates: First submitted 2021-01-09; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- viscotrabeculotomy (VT)). (Active Comparator)
  Interventions: Procedure: viscotrabeculotomy (VT)
- visco-circumferential-suture-trabeculotomy (VCST) (Active Comparator)
  Interventions: Procedure: visco-circumferential-suture-trabeculotomy (VCST) .
- Combined VT-Trabeculectomy with MMC (VT-Trab). (Active Comparator)
  Interventions: Procedure: combined VT-Trabeculectomy with MMC (VT-Trab).

INTERVENTIONS:
Procedure: viscotrabeculotomy (VT) — viscotrabeculotomy (VT)
  Arms: viscotrabeculotomy (VT)).
Procedure: visco-circumferential-suture-trabeculotomy (VCST) . — visco-circumferential-suture-trabeculotomy (VCST)
  Arms: visco-circumferential-suture-trabeculotomy (VCST)
Procedure: combined VT-Trabeculectomy with MMC (VT-Trab). — combined VT-Trabeculectomy with MMC (VT-Trab).
  Arms: Combined VT-Trabeculectomy with MMC (VT-Trab).

SUMMARY:
The current study aimed to compare between the long-term surgical outcomes of 3 surgical options (viscotrabeculotomy (VT), visco-circumferential-suture-trabeculotomy (VCST) or combined VT-Trabeculectomy with MMC (VT-Trab) in treatment of infants with (Primary Congenital Glaucoma (PCG)) below 1 month of age.

DETAILED DESCRIPTION:
This is a prospective, randomised controlled trial. We plan to recruit 60 infants with primary congenital glaucoma and younger than 1 month of age at the outpatient clinic of Mansoura Ophthalmic Center of Mansoura University in Mansoura, Egypt. Eyes will be randomly assigned to undergo one of 3 surgical interventions: viscotrabeculotomy (VT), visco-circumferential-suture-trabeculotomy (VCST) or combined VT-Trabeculectomy with MMC (VT-Trab).

The primary outcome of this study is compare the success rate in lowering IOP between the 3 surgical options in infants with Primary Congenital Glaucoma (PCG) below 1 month of age. The secondary clinical outcomes will include Intraocular pressure (IOP), horizontal corneal diameter, axial length, cup-disc ratio, refractive error and postoperative complications in these 3 surgical procedures. Data will be analysed. Complete success was defined as an IOP from 5 to 16 mmHg (under general anesthesia), without antiglaucoma drugs (AGD) or further surgical interventions, without progression of corneal diameter or disk cupping, and without serious visual complications. Qualified success was defined as fulfilling the same criteria but with the use of AGD.

ELIGIBILITY:
Inclusion Criteria:

Primary Congenital Glaucoma in Neonates

Exclusion Criteria:

secondary Congenital Glaucoma in Neonates. Congenital Glaucoma presented after 1 month of age.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
success rate in lowering intraocular pressure (IOP) | 3 years
  Complete success was defined as an IOP from 5 to 16 mmHg (under general anesthesia), without AGD or further surgical interventions, without progression of corneal diameter or disk cupping, and without serious visual complications. Qualified success was defined as fulfilling the same criteria but with the use of AGD.

SECONDARY OUTCOMES:
horizontal corneal diameter | 3 years
  The change in "white to white" corneal diameters in mm measured by caliber.
axial length | 3 years
  The change in axial length in mm measured by ultrasonography.
cup-disc ratio | 3 years
  The change in cup -disc ratio as measured by optical coherence tomography.
refractive error | 3 years
  The change in refractive error as measured by autorefractometer..

IPD SHARING:
Plan to Share IPD: Yes
providing data as supplemental digital content
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code